CLINICAL TRIAL: NCT00228527
Title: A Phase III, Multicentre, Randomized, Double-blind Parallel-group Study to Evaluate the Safety and Clinical Outcome of Once Daily Esomeprazole for the Treatment of Gastroesophageal Reflux Disease (GERD) in Pediatric Patients 1 to 11 Years of Age, Inclusive.
Brief Title: Esomeprazole for Treatment of GERD in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9614C00097
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Erosive Esophagitis; Non-erosive Esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole (Nexium)

SUMMARY:
To look at the safety and improvement in symptoms of a once a day dosing of esomeprazole in children 1 to 11 years old with inflammation of their esophagus or food pipe ("esophagitis") caused by gastroesophageal reflux disease (GERD) and diagnosed by endoscopy.

To verify the healing of the esophageal inflammation if the endoscopy reveals cuts in the lining of the food pipe.

To collect information that will describe the psychological, social, and economic effects on the primary caregiver of raising children ages 1 to 5 years old with GERD.

ELIGIBILITY:
Inclusion Criteria:

* Patients' parents/guardians must provide written informed consent prior to the execution of any study-related procedures.
* Patients who are able to comprehend their involvement in a clinical study, including risks and benefits, (typically ≥6 years of age) must have assent documented by study personnel prior to any study-related procedures.
* Patients must be diagnosed with endoscopically proven GERD by the investigator during the screening period or have a previous (within 2 weeks prior to Visit 1) diagnosis of erosive esophagitis by endoscopy and are candidates for PPI therapy.

Exclusion Criteria:

* Patients who have used a proton pump inhibitor within 14 days prior to randomization, including over-the-counter omeprazole.
* Patients who have used any prescription or over-the-counter (OTC) treatment (other than proton pump inhibitors) for symptoms of GERD, such as histamine 2 receptor antagonists or prokinetics, within 72 hours prior to randomization.
* Patients with a known hypersensitivity, allergy, or intolerance to any component of esomeprazole or omeprazole.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2004-10; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the safety of once daily treatment with esomeprazole in relieving GERD-associated symptoms in pediatric patients 1 to 11 years of age, inclusive.
The primary outcome variables include assessment of changes from baseline in medical history, physical examination, clinical laboratory evaluations, and adverse events.

SECONDARY OUTCOMES:
The secondary objective of the study is to evaluate the clinical outcome of once daily treatment with esomeprazole in relieving GERD-associated signs and symptoms in pediatric patients 1 to 11 years of age, inclusive.
The secondary objectives include:
- Assessment of changes from baseline in daily patient symptom assessment as reported by parent/guardian.
- Assessment of changes from baseline in Physician's Global Assessment
- Assessment of endoscopic healing of erosive esophagitis

CONTACTS AND LOCATIONS:
Locations (36):
- United States (24):
  - Research Site, Mobile, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Wilmington, Delaware
  - Research Site, Orlando, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Morristown, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, West Islip, New York
  - Research Site, Columbus, Ohio
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Norfolk, Virginia
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Brussels (Jette)
  - Research Site, Brussels (Laeken)
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Leuven
- France (3):
  - Research Site, Lille
  - Research Site, Paris
  - Research Site, Tours
- Italy (4):
  - Research Site, Genova, GE
  - Research Site, Parma, PR
  - Research Site, Roma, RM
  - Research Site, Napoli

REFERENCES:
- [Derived] Tolia V, Gilger MA, Barker PN, Illueca M. Healing of Erosive Esophagitis and Improvement of Symptoms of Gastroesophageal Reflux Disease After Esomeprazole Treatment in Children 12 to 36 Months Old. J Pediatr Gastroenterol Nutr. 2015 Jul;60 Suppl 1:S31-6. doi: 10.1097/MPG.0b013e3181ddcf11. PMID 26422096
- [Derived] Tolia V, Youssef NN, Gilger MA, Traxler B, Illueca M. Esomeprazole for the Treatment of Erosive Esophagitis in Children: An International, Multicenter, Randomized, Parallel-Group, Double-Blind (for Dose) Study. J Pediatr Gastroenterol Nutr. 2015 Jul;60 Suppl 1:S24-30. doi: 10.1097/01.mpg.0000469419.29000.94. PMID 26422095
- [Derived] Tolia V, Gilger MA, Barker PN, Illueca M. Healing of Erosive Esophagitis and Improvement of Symptoms of Gastroesophageal Reflux Disease After Esomeprazole Treatment in Children 12 to 36 Months Old. J Pediatr Gastroenterol Nutr. 2015 Jul;60 Suppl 1:S31-6. doi: 10.1097/MPG.0b013e3181ddcf11. PMID 26121348
- [Derived] Tolia V, Youssef NN, Gilger MA, Traxler B, Illueca M. Esomeprazole for the Treatment of Erosive Esophagitis in Children: An International, Multicenter, Randomized, Parallel-Group, Double-Blind (for Dose) Study. J Pediatr Gastroenterol Nutr. 2015 Jul;60 Suppl 1:S24-30. doi: 10.1097/01.mpg.0000469419.29000.94. PMID 26121347
- [Derived] Tolia V, Gilger MA, Barker PN, Illueca M. Healing of erosive esophagitis and improvement of symptoms of gastroesophageal reflux disease after esomeprazole treatment in children 12 to 36 months old. J Pediatr Gastroenterol Nutr. 2010 Nov;51(5):593-8. doi: 10.1097/MPG.0b013e3181ddcf11. PMID 20706150
- [Derived] Tolia V, Youssef NN, Gilger MA, Traxler B, Illueca M. Esomeprazole for the treatment of erosive esophagitis in children: an international, multicenter, randomized, parallel-group, double-blind (for dose) study. BMC Pediatr. 2010 Jun 11;10:41. doi: 10.1186/1471-2431-10-41. PMID 20540767
- [Derived] Gilger MA, Tolia V, Vandenplas Y, Youssef NN, Traxler B, Illueca M. Safety and tolerability of esomeprazole in children with gastroesophageal reflux disease. J Pediatr Gastroenterol Nutr. 2008 May;46(5):524-33. doi: 10.1097/MPG.0b013e318176b2cb. PMID 18493207